CLINICAL TRIAL: NCT00716235
Title: Characterization of Executive Functions and Patterns of Eye Movements in Children With Developmental Disabilities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Lidia Gabis, Sheba Medical Center
Other Study IDs: SHEBA-08-5185-LG-CTIL
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Attention Deficit Hyperactivity Disorder; Autistic Disorder; Developmental Coordination Disorder
Keywords: ADHD; ASD; PDD; DCD; Executive Functions
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autistic Disorder; Motor Skills Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- DCD: Children with a diagnosis of DCD
- Autism: Children with a diagnosis of Autism disorder
- ADHD: Children with a diagnosis of ADHD
- Control: Control group - children with no neurological or psychiatric problems

SUMMARY:
The purpose of this study is to characterize the profile of executive functions and eye movements in several populations of children with developmental disabilities.

DETAILED DESCRIPTION:
Abnormal Executive function (EF) profile was considered a major characteristic of Attention deficit / hyperactivity disorder (ADHD) and autism, and is frequently implicated in Developmental coordination disorder (DCD) children as well. The scientific literature implies that the EF profile among these three groups share some common abnormalities, but differ significantly in specific features. Abnormal EF profile may be a core feature of the developmental trajectory of each syndrome.

The fine measurement of eye movements may shed light on the underlying mechanisms of specific disorders, and point to abnormal attention, information processing, or motor organization. Gaze is an important component of social interaction. Eye contact and recognition of other's gaze direction are crucial to empathy assessment.

The current study will embark in the assessment of a wide range of EF in these populations and in a matched control group, as well as their relation to other important parameters such as daily function skills and comorbid neurobehavioral characteristics. It will also assess the pattern of eye movements in response to various visual stimuli in these populations. The main purpose is to characterize the similarities and differences of each of these populations, in terms of EF and eye movements.

Assessment methods:

Clinical parameters:

* Intelligence tests (according to the child's age)
* Communication: DSM-IV, ADOS, Stony Brook questionnaire
* Motor / Coordination: Movement Advanced Battery for Children (M-ABC)
* Attention: Conners Rating Scales - Revised (CRS-R 3rd ed.)
* Sleep: Sleep habits questionnaire

Executive functions will be assessed using the following methods:

* NEPSI-II
* BRIEF questionnaire
* Wisconsin Card Sorting Test
* Tower of Hanoi

Eye movements will be measured using an infra-red video camera produced by ISCAN inc. the following visual stimuli will be presented:

* Human faces presenting various emotions
* Various objects
* Saccade and anti-saccade tasks

ELIGIBILITY:
Inclusion Criteria:

* Age of 4-10 years
* A medical diagnosis according to the relevant study group
* Normal vision without glasses or contact lens.

Exclusion Criteria - clinical groups:

* Intelligence Quotient below 70
* A known brain damage
* A known hearing impairment
* Regular use of medications (except for psychostimulants)
* Evidence for a known genetic syndrome
* History of fetal CMV infection, birth asphyxia, major head injury or epilepsy

Exclusion Criteria - control group:

* Intelligence Quotient below 70
* Regular use of medications
* Evidence for a neurological / psychiatric disorder, birth injury, developmental delay, head injury, or other medical disorders that affect the central nervous system
* Family History - first degree) of autism, DCD, ADHD or other neurological/psychiatric disorder

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Gabis, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Weinberg Child Development Center, Sheba Medical Center, Tel-Hashomer, Ramat Gan, Israel

REFERENCES:
- See also: ISCAN Inc. - producing the eye tracking equipment for the study — http://www.iscaninc.com/